CLINICAL TRIAL: NCT01917383
Title: A Phase II Multi-center, Randomized Study to Evaluate the Monocular Addition of Trabodenoson (INO-8875) Ophthalmic Formulation to Latanoprost Ophthalmic Solution Therapy in Adults With Ocular Hypertension or Primary Open-Angle Glaucoma
Brief Title: A Phase II Study to Evaluate the Additivity of Trabodenoson to Latanoprost in Adults With Ocular Hypertension or Primary Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPC-01-2013
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Primary Open-Angle Glaucoma (POAG); Ocular Hypertension (OHT)
Keywords: glaucoma; primary open angle glaucoma; ocular hypertension; adenosine agonist; eye drop; trabodenoson; trabecular meshwork
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — trabodenoson; INO-8875; Latanoprost; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabodenoson Plus Latanoprost (Experimental): Experimental ophthalmic eye drop plus a prostaglandin analogue eye drop
  Interventions: Drug: Trabodenoson; Drug: Latanoprost
- Timolol Plus Latanoprost (Active Comparator): A Beta-blocker eye drop plus a prostaglandin analogue eye drop
  Interventions: Drug: Latanoprost; Drug: Timolol

INTERVENTIONS:
Drug: Trabodenoson — Ophthalmic eye drop
  Other Names: INO-8875
  Arms: Trabodenoson Plus Latanoprost
Drug: Latanoprost — Ophthalmic eye drop
  Other Names: Xalatan
Drug: Timolol — Ophthalmic eye drop
  Other Names: Timoptic
  Arms: Timolol Plus Latanoprost

SUMMARY:
The purpose of this study is to evaluate the intraocular pressure (IOP) lowering efficacy and the safety and tolerability profile of trabodenoson ophthalmic formulation compared to timolol maleate ophthalmic solution 0.5% in adults with ocular hypertension (OHT) or primary open-angle glaucoma (POAG) who are already receiving treatment with latanoprost ophthalmic solution 0.005% once every evening (QPM).

DETAILED DESCRIPTION:
Criteria

Inclusion Criteria:

1. Subject has signed and dated the current informed consent form (ICF).
2. Subject has the diagnosis of ocular hypertension (OHT) or primary open-angle glaucoma (POAG) (excluding secondary, pseudo-exfoliation, and pigment dispersion glaucomas).
3. Aged 18 or older.
4. Mean intraocular pressure (IOP) of ≥24 and ≤34 mm Hg.

Exclusion Criteria:

1. No significant visual field loss or any new field loss within the past year.
2. Cup-to-disc ratio ≥0.8
3. Central corneal thickness <500 µm or >600 µm
4. A recent (acute) or chronic medical condition that might obfuscate the Subject's study data

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated the current informed consent form (ICF).
2. Subject has the diagnosis of ocular hypertension (OHT) or primary open-angle glaucoma (POAG) (excluding secondary, pseudo-exfoliation, and pigment dispersion glaucomas).
3. Aged 18 or older.
4. Mean intraocular pressure (IOP) of ≥24 and ≤34 mm Hg.

Exclusion Criteria:

1. No significant visual field loss or any new field loss within the past year.
2. Cup-to-disc ratio ≥0.8
3. Central corneal thickness <500 µm or >600 µm
4. A recent (acute) or chronic medical condition that might obfuscate the Subject's study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chiltern, Bristol, Tennessee, United States